Efficacy of Psychological Intervention in Children with Cancer: A Randomized Controlled Trial (RCT) 14-August-2024

# SUMMARY OF PROCEDURES & STATISTICAL ANALYSIS PLAN

- 1. The study will be conducted at the Pediatric Oncology Unit of the Children's Hospital, PIMS Islamabad.
- 2. The study will involve 80 children aged 8-13 years who have been diagnosed with malignancies and are receiving chemotherapy.
- 3. Newly diagnosed pediatric cancer patients aged 8-13 years
- 4. Children must be receiving chemotherapy as part of their treatment plan.
- 5. Ability to participate in CBT sessions and complete assessment scales.
- 6. Single-blinded, two-arm randomized controlled trial (RCT).
- 7. **Experimental Group:** Receives five weekly sessions of Cognitive Behavioral Therapy (CBT).
- 8. **Control Group:** Receives usual care (UC), which includes standard medical and psychological support provided by the oncology unit.
- 9. Potential participants are identified by the oncology healthcare team at the time of cancer diagnosis.
- 10. Parents or guardians of eligible children are approached for consent, and assent is obtained from the children.
- 11. Randomization occurs immediately after enrollment.
- 12. Participants are randomly assigned to either the experimental group (CBT) or the control group (UC).
- 13. Randomization is conducted using a computer-generated random number sequence to ensure unbiased allocation.

- 14. **Allocation Concealment:** Allocation is concealed from the participants and the healthcare providers administering the usual care to minimize bias. However, the psychologist administering CBT cannot be blinded to group allocation.
- 15. Baseline assessments are conducted **immediately after** randomization and before any intervention begins.
- 16. Revised Child Anxiety and Depression Scale (RCADS): Used to assess levels of anxiety and depression in the children.
- 17. Pediatric Quality of Life Inventory (PedsQL) Generic Core Score 4.0: Used to assess the quality of life.
- 18. A trained psychologist or researcher administers the scales to the children.
- 19. The baseline assessment data provide a reference point for comparing post-intervention outcomes.
- 20. The CBT intervention begins immediately after the baseline assessment for those in the experimental group.
- 21. The CBT consists of five weekly sessions.
- 22. Duration: Each session lasts 30-35 minutes.
- 23. Content: The sessions focus on cognitive restructuring, relaxation techniques, coping strategies, and problem-solving skills tailored to the child's age and psychological needs.
- 24. Control Group: Children in the control group continue to receive usual care without any additional psychological intervention.
- 25. The endline assessment is conducted **one month after the** completion of the CBT intervention.

- 26. For participants in the experimental group, this is typically six weeks after baseline (allowing for five weeks of intervention and one-week post-intervention).
- 27. The same timeline applies to the control group, with the endline assessment conducted at a comparable time point.
- 28. The same trained psychologist or researcher who conducted the baseline assessment will administer the endline assessments to ensure consistency.
- 29. The primary outcomes (anxiety, depression, and quality of life) will be compared between the experimental and control groups using statistical methods appropriate for RCTs (e.g., ANCOVA adjusting for baseline values).
- 30. The analysis will determine whether the CBT intervention significantly reduces anxiety and depression and improves quality of life compared to usual care.

# Variables Typically Collected in an RCT for CBT Intervention in Pediatric Oncology Patients

#### 1. Demographic and Baseline Characteristics:

- Age: Continuous variable (years).
- Gender: Categorical variable (Male, Female).
- Type of Malignancy: Categorical variable (e.g., Leukemia, Lymphoma, Solid Tumor).
- **Stage of Cancer:** Categorical variable (e.g., Early, Intermediate, Advanced).
- Baseline Anxiety Score: Continuous variable, measured by RCADS.
- Baseline Depression Score: Continuous variable, measured by RCADS.
- Baseline Quality of Life (QoL) Score: Continuous variable, measured by PedsQL.

#### 2. Intervention-Related Variables:

- **Group Assignment:** Categorical variable (CBT Intervention, Usual Care).
- Attendance of CBT Sessions: Categorical variable (Number of sessions attended).
- Adherence to Usual Care: Categorical variable (Yes, No).

#### 3. Outcome Variables:

- Post-Intervention Anxiety Score: Continuous variable, measured by RCADS.
- Post-Intervention Depression Score: Continuous variable, measured by RCADS.
- Post-Intervention Quality of Life (QoL) Score: Continuous variable, measured by PedsQL.

#### 4. Additional Variables:

- Dropout Rate: Categorical variable (Yes, No).
- Adverse Events: Categorical variable (None, Mild, Moderate, Severe).

## **Baseline Characteristics Table:**

| Variable | CBT Group | Usual Care Group | p- |
|------------------------|-----------|------------------|-------|
| | (n=40) | (n=40) | value |
| Age (years, mean ± SD) | | | |
| Gender, n (%) | | | |
| Male | | | |
| -Female | | | |
| Type of Malignancy, n | | | |
| (%) | | | |
| - Leukemia | | | |
| - Lymphoma | | | |
| - Solid Tumor | | | |
| Stage of Cancer, n (%) | | | |
| - Early | | | |
| - Intermediate | | | |
| - Advanced | | | |
| Baseline Anxiety Score | | | |
| Baseline Depression | | | |
| Score | | | |
| Baseline QoL Score | | | |

#### **Post-Intervention Outcome Table:**

| Outcome | CBT Group | Usual Care Group | p- |
|-----------------------------|-----------|------------------|-------|
| | (n=40) | (n=40) | value |
| Post-Intervention Anxiety | | | |
| Score | | | |
| Post-Intervention | | | |
| Depression Score | | | |
| Post-Intervention QoL Score | | | |
| Dropout Rate, n (%) | | | |
| Adverse Events, n (%) | | | |
| - None | | | |
| - Mild | | | |
| - Moderate | | | |
| - Severe | | | |

## 3. Adherence and Session Attendance Table (for CBT Group Only)

| Variable | CBT Group | Usual Care Group |
|----------|-----------|------------------|
| | (n=40) | (n=40) |

| Attendance of CBT Sessions |
|--------------------------------|
| (mean ± SD) |
| Adherence to Usual Care, n (%) |